CLINICAL TRIAL: NCT07126860
Title: ZMoveMent-1: Effect of a Resistance and Aerobic Training Intervention on Quality of Life, Fitness, Immunological Parameters, and Oncological Outcome in Patients With Prostate Cancer
Brief Title: The Effect of a Structured Strength and Endurance Training Program on Quality of Life, Fitness, Blood Parameters and Survival in Prostate Cancer Patients
Acronym: ZMoveMent-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Shimon Kempin, Principal Investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-0573
Record Dates: First submitted 2025-07-31; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Metastatic Prostate Cancer; Prostate Cancer (Post Prostatectomy); Prostate Cancer Patients Treated by Radiotherapy; Prostate Cancer Non-Metastatic
Keywords: biomarkers; cardiovascular health; depression reduction; endurance training; resistance training; strength training; aerobic training; exercise intervention; fitness tests; functional capacity; mental health; muscle strength; physical activity; physical rehabilitation; prostate cancer; androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms; Psychological Well-Being; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Training (Experimental): The 12-week intervention phase comprises the initial 12 weeks of a home-based combined resistance and aerobic training protocol for the intervention arm. Training will commence 8 weeks (when medically cleared, a reduction to minimally 4 weeks is possible) after RP or completion of EBRT, or any time for PC patients undergoing systemic treatment. As part of their visit for baseline testing, participants will be familiarized with the online platform incorporating the training program, including the correct execution of the exercises. In addition, the online platform includes demonstration videos of all exercises.
  Interventions: Behavioral: Structured combined resistance and aerobic training
- Standard of Care (Other): The control arm will receive SOC, as well as a booklet with general information and guidelines about physical activity in prostate cancer patients, but without any specific exercise prescriptions.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Structured combined resistance and aerobic training — The 12-week intervention phase comprises the initial 12 weeks of a home-based combined resistance and aerobic training protocol for the intervention arm. Training will commence 8 weeks (when medically cleared, a reduction to minimally 4 weeks is possible) after RP or completion of EBRT, or any time for PC patients undergoing systemic treatment. As part of their visit for baseline testing, participants will be familiarized with the online platform incorporating the training program, including the correct execution of the exercises. In addition, the online platform includes demonstration videos of all exercises.
  Detailed information about the training program will be available for patients and investigators via a website and smartphone application. Additionally, participants will receive a printed document explaining the training program, the repetitions in reserve (RIR) scale (Helms et al., 2016), and the online tool/app for tracking.
  Arms: Structured Training
Behavioral: Standard of Care — Participants randomized to the SOC arm will also be informed about the benefits of exercise and motivated to engage in exercise under their own management (self-directed exercise). They will receive a booklet with general information and guidelines about physical activity in prostate cancer patients, but without any specific exercise prescriptions.
  Arms: Standard of Care

SUMMARY:
Prostate cancer is the second most common cancer among men. Many patients experience a significantly reduced quality of life due to either the cancer itself or the side effects of treatment. These side effects can include tiredness, weight gain, loss of muscle and strength, bone weakness, depression, reduced sexual function, and increased risk of heart problems. A commonly used treatment called androgen deprivation therapy, which reduces the levels of male hormones, can make these symptoms worse.

Previous research has shown that physical exercise-both strength training and endurance training-can help improve physical and mental well-being in men with prostate cancer. Regular exercise has also been shown to improve body composition, cardiovascular health, and reduce cancer-related fatigue. Some studies even suggest that exercise might support the immune system and slow down the progression of cancer.

The aim of this clinical trial is to find out whether a specific combination of resistance and aerobic training can help improve quality of life and health outcomes in men with prostate cancer. The exercise program is designed to be performed at home using simple equipment like resistance bands and bodyweight exercises, along with high-intensity interval training for endurance. Participants are asked to train three to six days a week.

150 men with prostate cancer at various stages of the disease will be included. These men will be randomly divided into two groups: two-thirds will receive the exercise program (intervention group), and one-third will continue with their usual care without the program (control group). The initial training period lasts 12 weeks and will be repeated to ensure that all participants in the exercise group train for at least six months. After that, they will be encouraged to keep training on their own.

The main goal of the study is to see if the exercise program leads to improvements in quality of life, physical fitness, body composition, and markers of immune function. It will also be analyzed how well the participants stick to the program, whether a longer training period has more benefits, how physically active the participants are overall, and how the program might affect other health and cancer-related outcomes.

The underlying hypothesis is that a structured, home-based resistance and aerobic training program will improve quality of life, physical fitness, body composition, immune function, and possibly cancer-related outcomes in men with prostate cancer.

DETAILED DESCRIPTION:
This study is a two-arm open-label controlled trial that aims to investigate the effects of combined resistance and aerobic training on quality of life (QoL), body composition, fitness parameters, immunological parameters, and oncological outcomes in patients with prostate cancer (PC).

150 men will be recruited with either localized, locally advanced, or metastatic PC. Patients will be randomly assigned in a 2:1 ratio to either the intervention arm (guided home-based training) or the standard of care (SOC) arm (self-directed or no exercise). Prior to enrollment, participants will provide written informed consent, undergo clinical eligibility confirmation, and complete screening assessments. Owing to the already documented general health benefits of exercise in patients with PC, participants randomized to the SOC arm will be informed about the benefits of exercise as well, and will be motivated to engage in exercise under their own management (self-directed exercise). Changes in physical activity will be monitored in both groups.

This study will include a screening phase, a 12-week intervention phase, a post-12-week intervention phase, and a longer-term intervention phase.

During the screening phase (maximally 35 days prior to the first training session), participants will undergo assessments to determine their eligibility for the study. This involves evaluating inclusion and exclusion criteria, as well as data collection on demographics and tumor stage. To avoid bias and to ensure equal participation and motivation of participants from both the intervention and the SOC arm in the baseline tests, patient randomization will only take place after the baseline testing.

The 12-week intervention phase comprises the initial 12 weeks of a home-based combined resistance and aerobic training protocol for the intervention arm. Training will commence 8 weeks (when medically cleared, a reduction to minimally 4 weeks is possible) after radical prostatectomy (RP) or completion of external-beam radiotherapy (EBRT), or any time for PC patients undergoing systemic treatment. As part of their visit for baseline testing, participants will be familiarized with the online platform incorporating the training program, including the correct execution of the exercises. In addition, the online platform includes demonstration videos of all exercises. The control arm will receive SOC without any exercise prescriptions. Throughout the phase, participants' physical activity will be monitored using regular questionnaires and wearable device data. Efficacy evaluations will be conducted at baseline and after the 12-week intervention phase.

The post-12-week intervention phase will follow the 12-week intervention phase and will last for 1 year. Throughout this phase, QoL, oncological outcomes, laboratory parameters, as well as ongoing physical activity will be assessed periodically.

The longer-term intervention phase will begin 1 year after completion of the 12-week intervention phase, and will continue until one of the following events occurs: death, loss to follow-up or withdrawal of consent, or end of the study, whichever occurs first. Throughout this phase, oncological outcomes will be assessed periodically.

The study population will consist of men diagnosed with localized, locally advanced, or metastatic PC. Participants with localized or locally advanced PC may be enrolled pre- or post- RP, or at any point before, during, or after EBRT. Training will then commence 4-8 weeks after completion of RP or EBRT. Participants with locally advanced, non-metastatic, and metastatic PC under systemic treatment and not undergoing local curatively intended treatment can be enrolled at any time under any treatment.

All measurements will be assessed at baseline (maximally 14 days prior to the first training session) and after the 12-week intervention phase. Additionally, laboratory parameters, patient-reported outcome (PRO) assessments, and wearable data assessments will be repeated 3, 6, and 12 months after completion of the 12-week intervention phase.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have a histologically diagnosed adenocarcinoma of the prostate
2. Participant has to be ≥ 18 years of age
3. Participant must have either localized, locally advanced, or metastatic PC which has been treated or is planned to be treated either by RP, EBRT, androgen deprivation therapy (ADT), androgen receptor signaling inhibitor (ARSI), or any combination
4. Participant must understand and remember the training regimen
5. Participant must have a smartphone to connect a wearable device
6. Participant must have a smartphone or computer to access the online platform
7. Participant has to be able to speak, understand, and read German or English
8. Participant must sign an informed consent form (ICF)

Exclusion Criteria:

1. Cardiovascular/neurological/musculoskeletal comorbidities with contraindications for resistance or aerobic training
2. High risk of pathological fracture due to unstable bone metastases (note: patients with bone metastasis are generally eligible for participation in the study and program as long as there is no acute high risk of fracture)
3. Any condition for which it may not be in the best interest of the patient to participate in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Functional Assessment of Cancer Therapy - Prostate (FACT-P) Questionnaire Score | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  Range of 0-156 points. Higher points mean higher QoL.
Change from Baseline in Total Muscle Thickness (TMT) | Baseline and after 12-week intervention phase
  Muscle Thickness (MT) will be measured via ultrasound (linear head held perpendicular to the skin) at 4 sites (anterior and posterior upper arm, anterior and lateral thigh). For the primary outcome, the sum of those 4 sites will be used (TMT), but the separate results will also be reported.
  The measurement protocol used is adapted from Schoenfeld et al. (2019): https://doi.org/10.1249/MSS.0000000000001764
Change from Baseline in Serum Low-Density Lipoprotein (LDL) in milligrams/deciliter (mg/dl) | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase

SECONDARY OUTCOMES:
Change from baseline in the Metabolic Equivalent of Task (MET)-minutes/week as reported by the World Health Organization (WHO) Global Physical Activity Questionnaire (GPAC) Questionnaire Score | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  The amount of MET-minutes in each GPAQ physical activity category (work, transport, leisure) will be reported.
Change from Baseline in Blood Pressure (systolic and diastolic) | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Adherence to the training program | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  Adherence will be assessed using different methods:
  1. Analysis of training platform: percentage of completed training sessions out of the total prescribed sessions
  2. Questionnaire: how many times per week and for how long (weeks) was the training program performed?
Adverse Events by Questionnaire | After 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  AE (e.g., bone pain, path. skeletal fracture, musculoskeletal injury, joint pain, falls, muscle soreness) will be monitored via questionnaire, and incidence, severity, type, and attribution (exercise/disease) will be recorded as case report forms. CTCAE (Common Terminology Criteria for Adverse Events) will be used as the grading system for AE.
Change from Baseline in the Expanded Prostate Cancer Index Composite (EPIC) Questionnaire Subscale Scores | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  Every subscale (urinary, bowel, sexual, hormonal) can range from 0-100. Higher scores mean higher QoL.
Change from Baseline in the Short Form 36 (SF-36) Questionnaire Subscale Scores | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  Every subscale (physical functioning, role limitations due to physical health, role limitations due to emotional health, fatigue, emotional well-being, social functioning, pain, general health) can range from 0-100. Higher scores mean higher QoL.
Change from Baseline in the International Index of Erectile Function (IIEF) Questionnaire Score | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  Score can range from 1-30. Higher score means better QoL (less erectile dysfunction).
Change from Baseline in the Pittsburgh Sleep Quality Index (PSQI) Questionnaire Score | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  Score ranges from 0-21. Higher Score means worse sleep quality.
Change from Baseline in the Decision Regret Scale (DRS) Questionnaire Score | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  Score ranges from 0-100. Higher score means higher regret (worse outcome).
Change from baseline in bodyweight in kilograms (kg) | Baseline and after 12-week intervention phase
Change from baseline in body mass index (BMI) in kg/(m^2) | Baseline and after 12-week intervention phase
  To calculate BMI, body weight in kg and body height in centimeters (cm) will be measured.
Change from baseline in hip- and waist circumference in cm | Baseline and after 12-week intervention phase
Change from baseline in muscle thickness (MT) at anterior upper arm, posterior upper arm, anterior thigh, and lateral thigh | Baseline and after 12-week intervention phase
  Muscle Thickness will be measured via ultrasound (linear head held perpendicular to the skin) at 4 sites (anterior and posterior upper arm, anterior and lateral thigh). The measurement protocol used is adapted from Schoenfeld et al. (2019): https://doi.org/10.1249/MSS.0000000000001764
Change from baseline in Short Physical Performance Battery (SPPB) Test Score | Baseline and after 12-week intervention phase
  The following SPPB data will be reported:
  * Balance test score (range 0-4, higher score means better performance)
  * 4 m gait speed test: score (range 0-4, higher score means better performance) and absolute time (in seconds)
  * Chair rising test: score (range 0-4, higher score means better performance) and absolute time (in seconds)
  * Overall score (0-12, higher score means better performance)
Change from baseline in Timed Up And Go Test (TUGT) in seconds | Baseline and after 12-week intervention phase
Change from baseline in grip strength test in newton/kilograms | Baseline and after 12-week intervention phase
Change from baseline in resting heart rate (RHR) in beats per minute (bpm), measured by wearable device | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  The mean RHR over the previous 14 days prior to the patient visit, as measured by the wearable device, will be reported.
Change from baseline in daily step count in steps/day, measured by wearable device | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  The mean daily step count over the previous 14 days prior to the patient visit, as measured by the wearable device, will be reported.
Change from baseline in daily caloric expenditure by activity in calories/day, measured by wearable device | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  The mean daily caloric expenditure by activity over the previous 14 days prior to the patient visit, as measured by the wearable device, will be reported.
Change from baseline in daily sleep duration in hours (h), measured by wearable device | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
  The mean daily sleep duration over the previous 14 days prior to the patient visit, as measured by the wearable device, will be reported.
Change from baseline in blood glucose level in mg/dl | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood creatinine level in mg/dl | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood C-reactive protein (CRP) level in mg/dl | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood alcaline phosphatase (AP) level in units/liter (U/l) | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood lactate dehydrogenase (LDH) level in U/l | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood total cholesterole level in mg/dl | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood high-density lipoprotein (HDL) level in mg/dl | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood insulin-like growth factor (IGF-1) level in ng/ml | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood hemoglobin in grams/deciliter (g/dl) | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood white blood cell (WBC) count in giga/liter (G/l) | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood platelet count in G/l | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood prostate-specific antigen (PSA) level in ng/ml | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood testosterone level in ng/ml | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood sex-hormone binding globulin (SHBG) level in nanomole/liter (nmol/l) | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase
Change from baseline in blood interleukin-6 (IL-6) level in picogram/ml (pg/ml) | Baseline, after 12-week intervention phase and 3/6/12 months after completion of 12-week intervention phase

OTHER OUTCOMES:
Event-free survival | 5 years after completion of 12-week intervention phase
  Events are defined as any event, whatever occurs earlier: biochemical failure, local-regional recurrence, first occurrence of distant metastases, radiographic progression on any imaging method, death for any reason
Overall survival | 5 years after completion of 12-week intervention phase
  Defined as the time from randomization to death for any reason
Patients with curative therapy: time until biochemical failure, metastasis-free survival | 5 years after completion of 12-week intervention phase
Patients with systemic therapy: progression-free survival, defined as radiographic progression on any imaging method or death for any reason, whichever occurs earlier | 5 years after completion of 12-week intervention phase
Percentage of men without an event at 1, 2, 3, 4, and 5 years | 5 years after completion of 12-week intervention phase
Time to first occurrence of symptomatic skeletal event (SSE = documentation of palliative RT, new fractures, spinal cord compression, change in antineoplastic therapy, surgical therapy) | 5 years after completion of 12-week intervention phase
Participant's Evaluation of the Training Program | After 12-week intervention phase
  A questionnaire collects feedback on usability, technical issues, and perceived helpfulness of both the wearable fitness tracker and the online training platform. Additionally, it evaluates the feasibility and safety of independently performing the exercise program, the clarity of the instructional videos, and the likelihood of continuing or recommending the program in the future. Responses are given on Likert scales and include yes/no options for specific technical issues and general recommendations.
Effect of training duration on the efficacy endpoints (< 6 months vs. < 12 months vs. > 12 months) | After completion of post-12-week intervention phase

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Brookman-May, Professor, Dr. med., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Ludwig Maximilian University Hospital Campus Großhadern, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No